CLINICAL TRIAL: NCT01570153
Title: Biomarkers Plus Bioimpedance Vector Analysis to Predict Cardiorenal Syndrome Onset and Prognosis in Patients With Acutely Decompensated Heart Failure: Biomonitoring and Cardiorenal Syndrome in Heart Failure(BIONICS-HF) Trial
Brief Title: Biomonitoring and Cardiorenal Syndrome in Heart Failure(BIONICS-HF) Trial
Acronym: BIONICS-HF
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, James L. Januzzi, JANUZZI, JAMES L, MD CARDIOLOGY DIVISION CARDIAC UNIT ASSOCIATES DIRECTOR CARDIAC CARE UNIT, Massachusetts General Hospital
Other Study IDs: 2012P000312
Record Dates: First submitted 2012-03-22; First posted 2012-04-04 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Cardiorenal Syndrome; Acute Decompensated Heart Failure
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 ml sample of blood will be draw into a tube containing ethylenediaminetetraacetic acid, spun for 15 minutes, and aliquoted to freezer tubes for biomarker measurement following the completition of the trial
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ADHF patients

SUMMARY:
The purpose of this study is to evaluate the ability of a non-invasive monitor that measures how much fluid is in the body as well as various blood tests for their ability to predict worsening kidney function in patients with heart failure.

DETAILED DESCRIPTION:
Our specific aims are to:

1. Evaluate the individual and collective ability of pro-B type natriuretic peptide (NT-pro-BNP), soluble (s)ST2, neutrophil gelatinase-associated lipocalin (NGAL), and bioelectrical impedance vector analysis (BIVA) for predicting in-hospital worsening renal function (WRF) in patients evaluated in emergency department (ED)with acutely decompensated heart failure (ADHF)compared to a model of clinical variables alone.
2. Evaluate the individual and collective ability of NT-proBNP, sST2, NGAL, and BIVA for identifying the correct cause of in-hospital WRF in patients evaluated in the ED with ADHF.
3. Evaluate the individual and collective ability of NT-pro-BNP, sST2, NGAL, and BIVA for predicting outcomes (all-cause death, all-cause re-hospitalization, initiation of renal replacement therapy by 180 days) in patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea thought to be due to ADHF
* NYHA class III or IV symptoms

Exclusion Criteria:

* renal failure requiring renal replacement therapy rior to enrollment
* unable or unwilling to participate
* > 6 hours from first dose of intravenous diuretic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department of the Massachusetts General Hospital with complaints compatible with Acute Decompensated Heart Failure (ADHF)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the onset of Worsening renal function following admission | From beginning of hospitalization to a follow up of 60 days

SECONDARY OUTCOMES:
the initiation of renal replacement therapy | From beginning of hospitalization to a follow up of 60 days
all cause mortality | From beginning of hospitalization to a follow up of 60 days

CONTACTS AND LOCATIONS:
Overall Officials: James L Januzzi, MD, Principal Investigator — Cardiology Division/Cardiac Unit Associated Director Cardiac Care Unit
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Ospedale Sant'Andrea, Rome, Italy

REFERENCES:
- [Background] Anwaruddin S, Lloyd-Jones DM, Baggish A, Chen A, Krauser D, Tung R, Chae C, Januzzi JL Jr. Renal function, congestive heart failure, and amino-terminal pro-brain natriuretic peptide measurement: results from the ProBNP Investigation of Dyspnea in the Emergency Department (PRIDE) Study. J Am Coll Cardiol. 2006 Jan 3;47(1):91-7. doi: 10.1016/j.jacc.2005.08.051. Epub 2005 Dec 9. PMID 16386670
- [Background] Manzano-Fernandez S, Januzzi JL Jr, Boronat-Garcia M, Bonaque-Gonzalez JC, Truong QA, Pastor-Perez FJ, Munoz-Esparza C, Pastor P, Albaladejo-Oton MD, Casas T, Valdes M, Pascual-Figal DA. beta-trace protein and cystatin C as predictors of long-term outcomes in patients with acute heart failure. J Am Coll Cardiol. 2011 Feb 15;57(7):849-58. doi: 10.1016/j.jacc.2010.08.644. PMID 21310322
- [Background] van Kimmenade RR, Januzzi JL Jr, Baggish AL, Lainchbury JG, Bayes-Genis A, Richards AM, Pinto YM. Amino-terminal pro-brain natriuretic Peptide, renal function, and outcomes in acute heart failure: redefining the cardiorenal interaction? J Am Coll Cardiol. 2006 Oct 17;48(8):1621-7. doi: 10.1016/j.jacc.2006.06.056. Epub 2006 Sep 27. PMID 17045898
- [Background] van Kimmenade RR, Pinto Y, Januzzi JL Jr. When renal and cardiac insufficiencies intersect: is there a role for natriuretic peptide testing in the 'cardio-renal syndrome'? Eur Heart J. 2007 Dec;28(24):2960-1. doi: 10.1093/eurheartj/ehl399. Epub 2007 Nov 5. No abstract available. PMID 17984131
- [Background] Ronco C, McCullough PA, Anker SD, Anand I, Aspromonte N, Bagshaw SM, Bellomo R, Berl T, Bobek I, Cruz DN, Daliento L, Davenport A, Haapio M, Hillege H, House A, Katz NM, Maisel A, Mankad S, Zanco P, Mebazaa A, Palazzuoli A, Ronco F, Shaw A, Sheinfeld G, Soni S, Vescovo G, Zamperetti N, Ponikowski P. Cardiorenal syndromes: an executive summary from the consensus conference of the Acute Dialysis Quality Initiative (ADQI). Contrib Nephrol. 2010;165:54-67. doi: 10.1159/000313745. Epub 2010 Apr 20. PMID 20427956
- [Background] Tang WH, Mullens W. Cardiorenal syndrome in decompensated heart failure. Heart. 2010 Feb;96(4):255-60. doi: 10.1136/hrt.2009.166256. Epub 2009 Apr 27. PMID 19401280
- [Background] Dupont M, Shrestha K, Tang WH. Revisiting the cardio-renal hypothesis: the pivotal role of the kidney in congestive heart failure. Eur J Heart Fail. 2011 Aug;13(8):820-2. doi: 10.1093/eurjhf/hfr092. No abstract available. PMID 21791537
- [Background] Gottlieb SS, Abraham W, Butler J, Forman DE, Loh E, Massie BM, O'connor CM, Rich MW, Stevenson LW, Young J, Krumholz HM. The prognostic importance of different definitions of worsening renal function in congestive heart failure. J Card Fail. 2002 Jun;8(3):136-41. doi: 10.1054/jcaf.2002.125289. PMID 12140805
- [Background] Maisel AS, Mueller C, Fitzgerald R, Brikhan R, Hiestand BC, Iqbal N, Clopton P, van Veldhuisen DJ. Prognostic utility of plasma neutrophil gelatinase-associated lipocalin in patients with acute heart failure: the NGAL EvaLuation Along with B-type NaTriuretic Peptide in acutely decompensated heart failure (GALLANT) trial. Eur J Heart Fail. 2011 Aug;13(8):846-51. doi: 10.1093/eurjhf/hfr087. PMID 21791540
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Mullens W, Abrahams Z, Skouri HN, Francis GS, Taylor DO, Starling RC, Paganini E, Tang WH. Elevated intra-abdominal pressure in acute decompensated heart failure: a potential contributor to worsening renal function? J Am Coll Cardiol. 2008 Jan 22;51(3):300-6. doi: 10.1016/j.jacc.2007.09.043. PMID 18206740
- [Background] Shah RV, Chen-Tournoux AA, Picard MH, van Kimmenade RR, Januzzi JL. Serum levels of the interleukin-1 receptor family member ST2, cardiac structure and function, and long-term mortality in patients with acute dyspnea. Circ Heart Fail. 2009 Jul;2(4):311-9. doi: 10.1161/CIRCHEARTFAILURE.108.833707. Epub 2009 May 14. PMID 19808354
- [Background] Januzzi JL Jr, Peacock WF, Maisel AS, Chae CU, Jesse RL, Baggish AL, O'Donoghue M, Sakhuja R, Chen AA, van Kimmenade RR, Lewandrowski KB, Lloyd-Jones DM, Wu AH. Measurement of the interleukin family member ST2 in patients with acute dyspnea: results from the PRIDE (Pro-Brain Natriuretic Peptide Investigation of Dyspnea in the Emergency Department) study. J Am Coll Cardiol. 2007 Aug 14;50(7):607-13. doi: 10.1016/j.jacc.2007.05.014. Epub 2007 Jul 30. PMID 17692745
- [Background] Rehman SU, Martinez-Rumayor A, Mueller T, Januzzi JL Jr. Independent and incremental prognostic value of multimarker testing in acute dyspnea: results from the ProBNP Investigation of Dyspnea in the Emergency Department (PRIDE) study. Clin Chim Acta. 2008 Jun;392(1-2):41-5. doi: 10.1016/j.cca.2008.03.002. Epub 2008 Mar 13. PMID 18387360
- [Background] Rehman SU, Mueller T, Januzzi JL Jr. Characteristics of the novel interleukin family biomarker ST2 in patients with acute heart failure. J Am Coll Cardiol. 2008 Oct 28;52(18):1458-65. doi: 10.1016/j.jacc.2008.07.042. PMID 19017513
- [Background] Nickolas TL, O'Rourke MJ, Yang J, Sise ME, Canetta PA, Barasch N, Buchen C, Khan F, Mori K, Giglio J, Devarajan P, Barasch J. Sensitivity and specificity of a single emergency department measurement of urinary neutrophil gelatinase-associated lipocalin for diagnosing acute kidney injury. Ann Intern Med. 2008 Jun 3;148(11):810-9. doi: 10.7326/0003-4819-148-11-200806030-00003. PMID 18519927
- [Background] Singer E, Elger A, Elitok S, Kettritz R, Nickolas TL, Barasch J, Luft FC, Schmidt-Ott KM. Urinary neutrophil gelatinase-associated lipocalin distinguishes pre-renal from intrinsic renal failure and predicts outcomes. Kidney Int. 2011 Aug;80(4):405-14. doi: 10.1038/ki.2011.41. Epub 2011 Mar 16. PMID 21412214
- [Background] Piccoli A. Bioelectric impedance measurement for fluid status assessment. Contrib Nephrol. 2010;164:143-152. doi: 10.1159/000313727. Epub 2010 Apr 20. PMID 20428000
- [Background] Di Somma S, De Berardinis B, Bongiovanni C, Marino R, Ferri E, Alfei B. Use of BNP and bioimpedance to drive therapy in heart failure patients. Congest Heart Fail. 2010 Jul;16 Suppl 1:S56-61. doi: 10.1111/j.1751-7133.2010.00162.x. PMID 20653713
- [Background] Peacock Iv WF. Use of bioimpedance vector analysis in critically ill and cardiorenal patients. Contrib Nephrol. 2010;165:226-235. doi: 10.1159/000313762. Epub 2010 Apr 20. PMID 20427973
- [Background] Piccoli A, Pittoni G, Facco E, Favaro E, Pillon L. Relationship between central venous pressure and bioimpedance vector analysis in critically ill patients. Crit Care Med. 2000 Jan;28(1):132-7. doi: 10.1097/00003246-200001000-00022. PMID 10667512
- [Background] Parrinello G, Paterna S, Di Pasquale P, Torres D, Fatta A, Mezzero M, Scaglione R, Licata G. The usefulness of bioelectrical impedance analysis in differentiating dyspnea due to decompensated heart failure. J Card Fail. 2008 Oct;14(8):676-86. doi: 10.1016/j.cardfail.2008.04.005. Epub 2008 Jun 6. PMID 18926440